CLINICAL TRIAL: NCT05297487
Title: Evaluation of the Early Use of the Pressure Relaxer in the Respiratory Impairment of Patients With Amyotrophic Lateral Sclerosis: Multicenter Randomized Controlled Study.
Acronym: RELAX SLA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021/CHU/08
Record Dates: First submitted 2022-03-07; First posted 2022-03-28 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care associated with daily and early use of (IPPB) intermittent positive pressure breathing (Experimental)
  Interventions: Device: early use of intermittent positive pressure breathing
- standard care alone (No Intervention)

INTERVENTIONS:
Device: early use of intermittent positive pressure breathing — standard care associated with daily and early use of intermittent positive pressure breathing
  Arms: standard care associated with daily and early use of (IPPB) intermittent positive pressure breathing

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a rare and serious neurodegenerative disease causing degeneration of motor neurons. . It leads to a progressive paralysis of the muscles involved in voluntary motricity. In France, its incidence is 2.5/100,000 inhabitants per year.

The death of patients is mainly caused by a progressive attack of the respiratory muscles. Indeed, the thorax is no longer actively mobilized to the maximum amplitude, it will lose its flexibility. A restrictive syndrome sets in followed by alveolar hypoventilation. Bronchial congestion may be concomitant.

Management is then based on non-invasive ventilation (NIV). This step, which is difficult for patients to accept psychologically, must be delayed as much as possible. However, to date, there are no precise recommendations on preventing the appearance of this restrictive syndrome and on slowing down the deterioration of lung function in patients.

The pressure relaxer (RLX) is an instrumental aid allowing on the one hand to mobilize the thorax thanks to hyper insufflations, and on the other hand to increase the effectiveness of the cough. The use of this device in physiotherapy is part of the HAS recommendations to promote decluttering.

However, we believe that RLX in patients with ALS, through the pulmonary alveolar recruitment it induces, could be relevant at an earlier phase, for the prevention of the decline in pulmonary functions: the restrictive syndrome, bronchial congestion and alveolar hypoventilation. So ultimately, the quality of life and survival of these patients would be improved.

It is in this context that this multicenter randomized controlled study RELAX'SLA takes place in order to evaluate the effects of the early use of the pressure relaxer on the respiratory impairment of patients with ALS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (over 18 years old) with a diagnosis of ALS,
* - Patient who presents with an impairment of the strength of the inspiratory muscles corresponding to the degradation of the Measurement of the maximum inspiratory pressure (MIP) and/or of the inspiratory pressure during the maximum sniffle (SNIP):
* Decrease in SNIP or MIP by 10% of previous values (measured at the last follow-up visit to the center in its standard care)
* If it is his first consultation (no previous value) we will include patients if they have SNIP or MIP values <90% of the theoretical values provided by the spirometer measuring the pressures. The SNIPs and MIPs (+/-1 standard deviation) must be disturbed for inclusion of the patient.
* Patient not yet using RLX for lung recruitment or Patient using RLX only as a decluttering aid.
* Person affiliated or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Patient with advanced restrictive impairment = FVC<50% of theoretical values on inclusion
* Patient with proven alveolar hypoventilation or treated with non-invasive ventilation
* Patient already treated with RLX for pulmonary recruitment
* Persons referred to in Articles L1121-5 to L1121-8 of the CSP (corresponding to all protected persons: pregnant woman, parturient, breastfeeding mother, person deprived of liberty by judicial or administrative decision, minor, and person making object of a legal protection measure: guardianship or curatorship)
* Patient with a contraindication to the use of RLX (1):
* Pneumothorax
* Known intracranial hypertension
* Hemodynamic instability
* Facial or skull surgery <6 months
* Tracheoesophageal fistula
* Active bleeding
* Untreated active tuberculosis
* Rebellious Hiccup
* the history of known emphysematous or bullous pathologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
assess the early use of the intermittent positive pressure breathing combined with standard management slows down the deterioration of lung volumes in patients with ALS | EVERY 3 MONTHS DURING 24 MONTHS
  Comparison of changes in lung volumes between the two groups based on Forced Vital Capacity (FVC), measured by spirometry during a Functional Respiratory Test (LFE)

IPD SHARING:
Plan to Share IPD: Undecided